CLINICAL TRIAL: NCT00489684
Title: Investigation of the Effect of Opioids on Experimental Hyperalgesia in Oesophagus and Skin, and in an Ischemic Model of Musclepain. Including an Explorative Study of the Effect of Morphine on the Pain Processing in the Brain
Brief Title: Effect of Opioids on Experimental Hyperalgesia in Oesophagus, Skin and Muscles
Acronym: AEO-2007-01
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Professor Asbjørn Mohr Drewes, Gastroenterological Outpatients Clinic, Aalborg Hospital, Aalborg
Other Study IDs: 2007-001881-33
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples are collected to study the pharmacokinetic of the drugs
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is a multi-modal multi-tissue human experimental pain study in 24 healthy volunteers. The study is a randomized cross-over study. The effect of 2 opioids will be compared on pain stimuli in skin, muscle an oesophagus. Hyperalgesia will be induced in skin and oesophagus, to sensitize these tissues. The pain thresholds before and after opioid administration will be compared. The hypothesis is that the difference in effect of the opioids is more pronounced in the presence of hyperalgesia. As hyperalgesia is a common phenomenon the clinic, the findings in this study may lead to a better understanding of the treatment of pain. The study will include an explorative study of the effect of Morphine of pain processing in the brain, this will provide us with new insight in the effect of the opioids of pain processing in the brain.

DETAILED DESCRIPTION:
The study is a multi-modal multi-tissue human experimental pain study in 24 healthy volunteers. The study is a randomized cross-over study. The effect of 2 opioids, Oxycodone and Morphine will be compared on pain stimuli in skin, muscle an oesophagus. Hyperalgesia will be induced in skin by capsaicin and in oesophagus by a mixture of capsaicin and acid, to sensitize these tissues. The pain thresholds before and after opioid administration will be compared. The hypothesis is that the difference in effect of the opioids is more pronounced in the presence of hyperalgesia. As hyperalgesia is a common phenomenon the clinic, the findings in this study may lead to a better understanding of the treatment of pain. The study will include an explorative study of the effect of Morphine of pain processing in the brain, this will provide us with new insight in the effect of the opioids of pain processing in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years
* Signed informed concent
* Healthy
* Women must use a safe contraceptive method
* Negative pregnancy test

Exclusion Criteria:

* Pregnancy
* Allergy to study medication
* Participating in another medicine study
* Previous addictive behaviour
* Need for other treatments
* Use of strong analgesics
* Use of any analgesics 24 hours before the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-08; Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Mohr Drewes, Professor, Principal Investigator — Aalborg Hospital S. Gastroenterological Outpatients clinic
Locations (1):
- Gastroenterological outpatients clinic, Aalborg, Aalborg, Denmark